CLINICAL TRIAL: NCT02684539
Title: Autonomous Syncope Onset Prediction and Prevention An Open-label, One-centre Pilot Study on Healthy Subjects With the Erigo Tilt Table
Brief Title: Autonomous Syncope Onset Prediction and Prevention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: project weill not be realized for organisational reasons
Sponsor: Swiss Federal Institute of Technology (Other)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EF1
Record Dates: First submitted 2015-11-27; First posted 2016-02-18 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tilt table Erigo® (Experimental): observation of physiological parameters, tilting table with onset of syncope
  Interventions: Device: tilt table Erigo®

INTERVENTIONS:
Device: tilt table Erigo® — tilting table with onset of syncope

SUMMARY:
syncope prediction on tilt table

DETAILED DESCRIPTION:
A tilt table is used to provoke syncope. syncope prediction is achieved through sensor measurements (ECG, ICG, SpO2, breathing rate, BP, NIRS, GSR, oculography).

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

-

Ages: 18 Years to 49 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
clinical sign of syncope | 1 session of 90 minutes duration
  as diagnosed by the medical staff

IPD SHARING:
Plan to Share IPD: No